CLINICAL TRIAL: NCT06014541
Title: A Prospective and Retrospective Observational/Non-interventional Study to Characterize Biomarkers and Disease Progression in Patients With MECP2 Duplication Syndrome
Brief Title: Observational Study to Characterize Biomarkers and Disease Progression in Participants With Methyl CpG Binding Protein 2 (MECP2) Duplication Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NH00006
Record Dates: First submitted 2023-08-09; First posted 2023-08-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Methyl CpG Binding Protein 2 (MECP2) Duplication Syndrome
Keywords: MDS
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — CSF and blood samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MECP2 Duplication Syndrome Disease Participants: Participants with a diagnosis of MDS with genetic confirmation of MECP2 duplication (or triplication) will undergo CSF and blood collection, electrophysiological and clinical assessments, up to Week 104 as a part of prospective study. Each participant's medical and family history data will be collected retrospectively from available medical notes and charts, from birth up to the end of the study (up to 110 weeks). Participants will have an option to participate in an optional sub-study that will capture pre-defined list of activities at home video.

SUMMARY:
The purpose of the study is to prospectively assess longitudinal changes in biomarkers (MECP2, potential biomarkers of target engagement and disease activity) in cerebrospinal fluid (CSF) and blood; characterize longitudinal changes in performance on clinical scales (clinician-reported measures of neurodevelopment and functioning) and caregiver-reported outcome assessments (communication, gastrointestinal, social-emotional-adaptive behavioral measures); evaluate longitudinal changes in caregiver-reported health-related quality-of-life measures; and assess the frequency, type, and severity of seizures over time.

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, non-interventional prospective and retrospective study in up to 40 participants with MECP2 duplication syndrome (MDS) who can undergo general anesthesia or conscious sedation to collect fluid biomarkers (CSF and blood), undergo electrophysiological assessments (electroencephalogram [EEG], evoked potentials [EP], pupillometry), clinical assessments and caregiver reported outcomes measures, to be used in support of the development of therapies for MDS. The study duration for each participant will be approximately 110 weeks.

ELIGIBILITY:
Key Inclusion Criteria

* Participant has a diagnosis of MDS with genetic confirmation of MECP2 duplication (or triplication)
* Participant has a parent or caregiver (CG) ≥ 18 years old capable of providing informed consent (signed and dated), and able to attend all scheduled study visits and provide feedback regarding the participant's symptoms and performance as described in the protocol and be able to comply with all study requirements and activities
* Male ≥ 1 month and ≤ 65 years of age
* No contraindications for lumbar puncture (LP)'s, blood draws, sedation (if necessary) or other study activities
* Medically stable to complete the study and will tolerate sedation or general anesthesia and other study activities

Key Exclusion Criteria

* Clinically significant abnormalities in medical history (e.g., clinically significant renal, hepatic, or cardiac abnormalities; major surgery within 3 months of screening) or upon physical examination that could potentially impact the NH of MDS
* Unwillingness or inability to comply with study procedures, including follow up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator
* Treatment with an investigational drug, gene therapy, stem cell therapy, biological agent, or device within 30 days of screening, or 5 half-lives of investigational agent, whichever is longer (participants cannot be concurrently enrolled in NH00006 and ION440-CS1).

Ages: 1 Month to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male participants who have a diagnosis of MDS, with genetic confirmation of MECP2 duplication (or triplication) will be enrolled.
Study Population: Participants who have a diagnosis of MDS with genetic confirmation of MECP2 duplication or triplication will be enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in MeCP2 in the CSF | Baseline and on Weeks 13, 26, 39, 52
Laboratory biomarkers for MECP2 Duplication | Baseline and on Weeks 13, 26, 39, 52
  Proteomic analysis of plasma samples to determine biomarkers of disease progression.
Change From Baseline in MECP2 Duplication Syndrome Severity Scale Across All Domains | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in the Revised Motor Behavioral Assessment | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in the Bayley Scales of Infant and Toddler Development, 3rd Edition | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in Vineland Adaptive Behavior Scales 3rd Edition | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in Observer Reported Communication Ability Measure | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in Quality-of-Life Inventory-Disability Score | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in the Frequency of Seizures | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in Global Assessment of Severity of Epilepsy Scale Score | Baseline and on Weeks 13, 26, 39, 52, 78, 104

SECONDARY OUTCOMES:
Change From Baseline in Auditory Evoked Potential | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Change From Baseline in Visual Evoked Potentials | Baseline and on Weeks 13, 26, 39, 52, 78, 104
Perform a retrospective chart review of the participant's medical history and family history to characterize the natural history of MDS | Baseline and on Weeks 13, 26, 39, 52, 78, 104

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCSD - Rady Children's Hospital, San Diego, California
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No